CLINICAL TRIAL: NCT04654624
Title: Child Discomfort and Parental Acceptability of Silver Diamine Fluoride and Alternative Restorative Treatment: a Randomized Controlled Clinical Trial
Brief Title: Child Discomfort and Parental Acceptability of Silver Diamine Fluoride and Alternative Restorative Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other); Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDF vs. ART
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Dental Caries; Child Discomfort
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Diamine Fluoride (Experimental)
  Interventions: Drug: SDF
- Atraumatic Restorative Treatment (Active Comparator)
  Interventions: Drug: ART

INTERVENTIONS:
Drug: SDF — Steps of SDF 38% application were carried out following the manufacturer's instructions. Eligible primary carious teeth were first dried and isolated using cotton rolls and gauze. Adjacent soft tissues were isolated using petrolleum gelly in order to prevent any irritation or staining from SDF that was directly placed into the carious lesion using a microbrush, allowed to absorb for 2 minutes, then dried with air. Parents were instructed that children should not eat for one hour after treatment. The second application was done after 6 months.
  Arms: Silver Diamine Fluoride
Drug: ART — Steps of ART caries removal were carried out following the Frencken et al. criteria where the cavity opening was widened using the tip of a dental hatchet. The carious dentin was then removed using a spoon excavator starting at the enamel-dentin junction, unsupported enamel was removed using the hatchet, and finally the cavity was cleaned using a wet cotton pellet and dried. After complete removal of infected dentin, the cavity walls and floor were conditioned for 10 seconds, washed and dried with cotton pellets, then restored with chemically cured glass ionomer cement that was applied under finger pressure, then coated with petroleum jelly.
  Arms: Atraumatic Restorative Treatment

SUMMARY:
The aim of the current study was to compare pain perception of young children treated with SDF and ART, as well as their parents' acceptability of both modalities.

DETAILED DESCRIPTION:
Eighty, 3-8-years-old children, having at least one deciduous asymptomatic tooth with active caries were randomly assigned into 2 groups; SDF for caries arresting in the test group, and ART for caries removal in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Negative and definitely negative behavior according to Frankl's behavior rating scale.
* Having at least one deciduous asymptomatic tooth with active caries, as defined by the International Caries Detection and Assessment System; ICDAS II scores 4, 5, 6.

Exclusion Criteria:

* Children who suffered from silver allergy, oral ulcerations, pulpal infections and whose parents needed immediate permanent restorations.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Pain perception | 6 months
  Pain reaction was assessed using the Sound, Eye, Motor scale (SEM) according to Wright et al. criteria. It is an objective method for pain assessment, where the child's level of anxiety was evaluated according to three types of observations. The score in each category ranged from one (no pain) to four (intense pain). A lower score represents less physical reaction to the procedure than does a higher value. Time of treatment was recorded using a stopwatch.

SECONDARY OUTCOMES:
Parents' acceptability of the treatment modality | 2 weeks
  It was assessed using a 5-likert scale, self-administered questionnaire, specifically designed for the current study.

CONTACTS AND LOCATIONS:
Overall Officials: Amel M Ahmed, Phd, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt and College of Dentistry, Princess Nourah Bint Abdulrahman University, Riyadh, Saudi Arabia; Hoda M Abdellatif, PhD, Study Chair — College of Dentistry, Princess Nourah Bint Abdulrahman University, Riyadh, Saudi Arabia and College of Dentistry Texas A&M University, Texas, USA; Sarah I Baghdady, M.Sc, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Wafaa E Abdelaziz, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Mona A ElKateb, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt and College of Dentistry, Princess Nourah Bint Abdulrahman University, Riyadh, Saudi Arabia
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Wright GZ, Weinberger SJ, Marti R, Plotzke O. The effectiveness of infiltration anesthesia in the mandibular primary molar region. Pediatr Dent. 1991 Sep-Oct;13(5):278-83. PMID 1815200
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963